CLINICAL TRIAL: NCT00362999
Title: Histamine Pharmacodynamics in Patients With Allergic Rhinitis: Validation of Laser Doppler Flowmetry as a Surrogate Endpoint
Brief Title: Validation of Laser Doppler Flowmetry to Identify Allergic Rhinitis Patients With Pharmacogenetic Alterations in Histamine Metabolism
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Bridgette Jones, Associate Professor of Pediatrics, MD, MSCR, Children's Mercy Hospital Kansas City
Other Study IDs: 11120477
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Allergic Rhinitis
Keywords: Allergic; Rhinitis; Pharmacogenetics; Histamine
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis to be proven is that histamine iontophoresis with measurement of microvascular blood flow by laser Doppler flowmetry can be used as a reliable marker to characterize the normal microvascular cutaneous response to histamine.

DETAILED DESCRIPTION:
The specific aim of this study is to validate iontophoresis (with measurement of microvascular blood flow by laser Doppler flowmetry) in a pediatric cohort as a surrogate marker capable of reliably characterizing the normal physiologic response of the cutaneous microvasculature to histamine. In future studies laser Doppler flowmetry ultimately will be used to assess whether microvascular blood flow determined by a previously validated laser Doppler technique can be used as a reliable surrogate endpoint capable of functionally discriminating the effects of polymorphisms in the genes which are quantitatively important for histamine metabolism. The hypothesis to be proven is that histamine iontophoresis with measurement of microvascular blood flow by laser Doppler flowmetry can be used as a reliable marker to characterize the normal microvascular cutaneous response to histamine.

ELIGIBILITY:
Inclusion Criteria:

-Established diagnosis of allergic rhinitis and/or allergic conjunctivitis, and/or allergic asthma either clinically (by presence of rhinitis and/or conjunctivitis with or without associated wheezing) and/or with a positive RAST/skin test to the following allergens: trees, grass, weeds, molds, cat, dog, dust mites and/or cockroach)

Exclusion Criteria:

* Previous history or laboratory evidence of McCune Albright syndrome, immunodeficiency, mastocytosis, receipt of immunomodulatory treatment, chronic conditions associated with abnormalities of the integument, hepatic or renal compromise, neoplastic disease, movement or neurologic disorders and uncontrolled ADHD
* Active atopic dermatitis at the site of the skin prick test or site where histamine iontophoresis will be performed, i.e. active atopic dermatitis on anterior forearms
* History of anaphylaxis or anaphylactic like episode
* Evidence of pregnancy (by urinary hCG) or lactation
* Use of drugs (within a specified time period) of agents capable of altering the response to histamine provocation (e.g., antihistamines, systemic corticosteroids, tricyclic antidepressants)
* Presence of any condition that, in the opinion of the investigator, would produce difficulty with adherence to study procedures.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with allergic rhinitis
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2024-07 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
comparison of histamine iontophoresis laser doppler monitoring with epicutaneous histamine testing in measuring the microvasculature response to histamine | one time point

SECONDARY OUTCOMES:
intra-individual variability of histamine iontophoresis with laser doppler monitoring | at least 6 months
  Determine the intra-individual variability of histamine iontophoresis with laser doppler flowimetry.
  Twenty subjects will be asked to return for 2 more visits for histamine iontophoresis with laser doppler flowimetry and the intra-individual variability of the measurement will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette L Jones, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States